CLINICAL TRIAL: NCT04681768
Title: Abemaciclib in Combination With Endocrine Therapy as First Line Therapy in Metastatic Breast Cancer Patients With Symp-tomatic Visceral Metastases or High Tumor Burden
Brief Title: Abemaciclib in Combination With Endocrine Therapy as First Line Therapy in Metastatic Breast Cancer Patients
Acronym: Abemacare
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: I3Y-NS-O003
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer/ Metastatic Breast Cancer
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Correlation analyses between circulating tumor DNA (ctDNA), protein tumormarkers and ORR/CRR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib tablets 150 mg, 100 mg, 50 mg as clinical routine: 150 mg twice daily per os, in-label administration in combination with endocrine therapy (aromatase inhibitor or Fulvestrant)
  Other Names: Verzenios®

SUMMARY:
Breast cancer is one of the most common cancers in women. 20-30 % of all breast cancer patients are faced with advanced disease, comprising both locally advanced breast cancer (LABC) and metastatic breast cancer (MBC). 80% of MBC cases are diagnosed as hormone receptor (HR) positive disease. The main systemic treatment options for these women include endocrine therapy (ET). The need of over-coming de novo or acquired resistance to ET in metastatic breast cancer has led to the integration of CDK4/6 inhibitors into combined ET of MBC. Abemaciclib represents a selective and potent small molecule inhibitor of CDK4/6 which has been granted approval by the European Medical Association (EMA). In two phase III trials Abemaciclib has been shown to double treatment efficacy in terms of PFS prolongation, to improve ORR and to prolong overall survival. At the same time, it has been shown that side effects of the drug are well manageable and QoL of patients under Abemaciclib is maintained.

DETAILED DESCRIPTION:
Against the above discussed background there is a clear rationale to further collect real world data confirming that the use of endocrine based therapy in metastatic breast cancer is beneficial for the patient cohort with symptomatic visceral metastases and high tumor burden. Data recently presented, showed that Abemaciclib in combination with Letrozole leads to substantial reduction in tumor size after only two cycles of therapy. Since Abemaciclib is the only CDK4/6-inhibitor that can be given "steady state" without a "one-week-off"-period and since there has been beginning evidence that Abemaciclib is penetrating the blood brain barrier in patients with brain metastases, it seems reasonable to choose Abemaciclib in combination with endocrine therapy for an observational study whose objective will be to collect efficacy data within clinical routine on Abemaciclib in combination with endocrine therapy within a cohort of ERpos/HER2neg breast cancer patients with symptomatic visceral metastases or high tumor burden.

LDH-levels above 400 U/l as well as abnormal levels of breast cancer specific tumor markers CA 15-3 and CEA have been proven to correlate with disease extent in metastatic breast cancer and thus can be used to identify metastatic breast cancer patients with high tumor burden. Recently it could be shown that circulating tumor DNA (ctDNA) bares greater correlation with changes in tumor burden than CA 15-3 and can provide the earliest measure of treatment response in women with metastatic breast cancer. This warrants further research to evaluate ctDNA as a tool for measuring early tumor response in MBC patients.

Translational research part:

In the era of personalized cancer therapy, testing for genetic alterations has become an essential tool in clinical practice. It allows clinicians to identify patients who are most likely to benefit from molecularly targeted treatments. Currently, evaluation of response to targeted drugs is largely based on imaging (CT or MRT), an approach unable to reveal mechanistic details on individual treatment effects. Sequential biopsies of tumors and their molecular analysis could yield additional information, but repetitive sampling of tissue that is representative and adequate in quantity and quality is rarely feasible, especially in the metastatic disease setting.

Liquid biopsies (LBs) represent a minimally-invasive alternative of great potential in this setting. Although recent technical advances allow very sensitive detection of LB-based tumor biomarkers, only few LB assays have yet entered into clinical routine.

Blood plasma samples from patients treated with Abemaciclib will be analyzed to identify predictive cell-free (cf) DNA-based biomarkers as indicators for treatment efficacy and early detection of resistance. To this end, cfDNA will be screened for mutations using a targeted next-generation sequencing panel (AVENIO ctDNA Expanded Kit, Roche). This panel is covering a total of 192 kb and consists of 77 genes, including those currently in the US National Comprehensive Cancer Network guidelines as well as emerging biomarkers currently being investigated in clinical trials.

For each plasma sample, concentration of cfDNA as well as presence and allelic frequencies of tumor mutations will be measured. Additionally, associations with progression-free survival and overall survival will be evaluated using Cox regression models. Clinical variables will be used as covariates in multivariable regression models to evaluate the independence of the LB-based biomarkers.

As a result, the investigators hope to identify minimally invasive LB-based biomarkers for serial monitoring of metastatic breast cancer patients. These biomarkers could add to the prediction of therapy response as well as the early detection of therapy resistance towards endocrine therapy and Abemaciclib.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Female patients who will start endocrine therapy (aromatase inhibitor or Fulvestrant) in combination with Abemaciclib as first line treatment for metastatic breast cancer within clinical routine
3. Signed informed consent
4. Life expectancy greater or equal to 12 weeks
5. Histologically proven diagnosed estrogen receptor positive, HER2 negative metastatic breast cancer not amenable to curative treatment
6. Radiographic evidence of measurable or evaluable visceral disease
7. Visceral involvement must fulfil one of the following criteria:

   1. Presence of any clinical sign or symptom from visceral disease (at least one of the following: pleural effusion, ascites, abdominal pain from liver or peritoneal metastases, dyspnea from pleural effusion or lymphangiosis of the lung, elevated liver enzymes (> 2x ULN), elevated bil-irubin)
   2. Signs of high tumor burden (at least one of the following: LDH >399 U/l with K in normal range, abnormal (> 2x ULN) CEA or CA15-3 level, radiographic signs of lymphangiosis of the lung, cytologically proven bone marrow infiltration)

Exclusion Criteria:

1. Contraindications for treatment with Abemaciclib, aromatase inhibitor or Fulvestrant according to current SmPC
2. Prior first line therapy (endocrine or chemotherapy) for metastatic breast cancer
3. Prior treatment with any CDK4/6 inhibitor (or participation in any CDK4/6 inhibitor clinical trial for which treatment assignment is still blinded)
4. Bone-only disease
5. Participation in clinical trials using an IMP within the last four weeks prior to inclusion (ICF)
6. Treatment with a drug that has not received regulatory approval for any indication within 28 days of initiation of study treatment for a non-myelosuppressive or myelosuppressive agent, respectively
7. Patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer/ metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) while being on study treatment using RECIST V1.1. | Maximum time frame will be 48 months
  Aim of this observational study is to collect efficacy data within clinical routine on Abemaciclib in combi-nation with endocrine therapy in estrogen receptor (ER) positive, HER2 negative metastatic breast cancer patients with symptomatic visceral disease or disease with high tumor burden.

SECONDARY OUTCOMES:
ORR at first, second and third time point of tumor evaluation | Maximum time frame will be 48 months
  ORR at first, second and third time point of tumor evaluation (according to clinical routine every 8 weeks) defined as the proportion of patients with having partial or complete response at first, second and third time point of tumor evaluation after initiation of study treatment using RECIST V1.1.
Disease control rate (DCR= CR+PR+SD) at first, second and third time point of tumor evaluation | Maximum time frame will be 48 months
  Disease control rate (DCR= CR+PR+SD) at first, second and third time point of tumor evaluation after initiation of study treatment (according to clinical routine every 8 weeks)
Duration of response (DoR) | Maximum time frame will be 48 months
  Duration of response (DoR), defined as the time from first documentation of OR to first documentation of PD according to RECISTV1.1 or death of any cause
Clinical response rate (CRR) at 4, 8, 16 and 24 weeks after initiation of study treatment | zp to 24 weeks
  Clinical response rate (CRR) at 4, 8, 16 and 24 weeks after initiation of study treatment defined as the proportion of patients assessed by the investigator as having at least one sign or symptom of clinical response.
Clinical benefit rate (CBR) | Maximum time frame will be 48 months
  Clinical benefit rate (CBR), defined as the percentage of patients with CR, PR or SD for at least 24 weeks [Time frame: initiation of study treatment to PD or death of any cause
Time to initial response (TTR) | Maximum time frame will be 48 months
  Time to initial response (TTR), defined as the time from initiation of study treatment to first documentation of objective response
Progression-free survival (PFS) | Maximum time frame will be 48 months
  Progression-free survival (PFS), defined as the time from initiation of study treatment until objective tumor progression or death, whichever occurs first
Time to treatment failure (TTF) | Maximum time frame will be 48 months
  Time to treatment failure (TTF), defined as the time from initiation of study treatment to discon-tinuation of treatment for any reason, including disease progression, treatment toxicity, and death
Change in tumor size | Maximum time frame will be 48 months
  Change in tumor size, defined as change of largest tumor-diameter on baseline tumor evaluation during the course of study treatment
Frequency of AE/SAE during study | Maximum time frame will be 48 months
  occurenec of AE/SAE during study
Patient reported outcomes (PRO) | Maximum time frame will be 48 months
  Patient reported outcomes (PRO): change from baseline to end of study in symptom burden and quality of life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Minimum score =0 Maximum score = 100. Higher score would mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ettl, MD, Study Chair — Klinikum rechts der Isar der TU München, Klinik und Poliklinik für Frauenheilkunde
Locations (1):
- Klinikum rechts der Isar der TU München, Klinik und Poliklinik für Frauenheilkunde, Munich, Germany

IPD SHARING:
Plan to Share IPD: No
it is not planed to share IPDs